CLINICAL TRIAL: NCT00128531
Title: Efficacy and Safety of a New Leuprolide Acetate 3.75 mg Depot Formulation, GP-Pharm S.A., When Given as Palliative Treatment to Prostate Cancer Patients
Brief Title: Leuprolide Acetate 3.75 mg Depot to Treat Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GP-Pharm (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRO-04-62
Record Dates: First submitted 2005-08-08; First posted 2005-08-10 (Estimated); Last update posted 2007-11-14 (Estimated); Status verified 2007-11

CONDITIONS: Prostate Cancer
Keywords: Phase III; open label; multiple dose; safety study; pharmacokinetic study; efficacy study
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide

INTERVENTIONS:
Drug: leuprolide acetate

SUMMARY:
The purpose of this study is to look at the efficacy and safety of leuprolide acetate in patients with prostate cancer.

DETAILED DESCRIPTION:
Other assessments include evaluation of main leuprolide PK parameters in 12 subjects after administration of 3 doses.

Study Design:

This will be a multi-center, open-label, fixed investigation of six monthly dosages of leuprolide acetate 3.75 mg administered to patients with histologically proven carcinoma of prostate, who might benefit from medical androgen deprivation therapy.

A total of 120 male patients will receive a single, i.m. injection of leuprolide acetate 3.75 mg initially on study day 0 (after baseline assessment) and then monthly (i.e. every 28 days) for five months.

12 of the patients will also have plasma leuprolide levels measured for PK analysis during the first 3 injection periods (PK group). These patients will belong to pre-defined study sites.

ELIGIBILITY:
Inclusion Criteria:

* Males >/= 18 years of age, with histologically proven carcinoma of the prostate, who might benefit from medical androgen deprivation therapy
* Life expectancy of at least 1 year
* World Health Organization/Eastern Cooperative Oncology Group (WHO/ECOG) performance status of 0, 1, or 2
* Adequate renal function at screening as defined by serum creatinine </= 1.6 times the ULN (upper limit of normal) for the clinical laboratory
* Adequate and stable hepatic function as defined by bilirubin </= 1.5 times the ULN and transaminases (i.e. SGOT, SGPT) </= 2.5 times the ULN for the clinical laboratory at screening
* Ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the Investigator and to comply with the requirements of the entire study
* Signed written informed consent prior to inclusion in the study

Exclusion Criteria:

* Evidence of brain metastases, in the opinion of the Investigator, taking into account medical history, clinical observations and symptoms
* Evidence of spinal cord compression, in the opinion of the Investigator, taking into account medical history, clinical observations and symptoms
* Evidence of severe urinary tract obstruction with threatening urinary retention, in the opinion of the Investigator, taking into account medical history, clinical observations and symptoms
* Excruciating, severe pain from extensive osseous deposits, in the opinion of the Investigator, taking into account medical history, clinical observations and symptoms
* Testosterone levels < 1.5 ng/mL at screening, locally determined at the laboratory of each clinical site
* Previous cancer systemic therapy such as chemotherapy, immunotherapy (e.g. antibody therapies, tumor-vaccines), biological response modifiers (e.g. cytokines) within 3 months of baseline
* Previous hormonal therapy for treatment of prostate cancer, such as luteinising hormone-releasing hormone (LHRH) analogues (e.g. Lupron®, Zoladex®, etc.) [no wash-out allowed]
* Previous treatment with androgen receptor (AR) blockers, such as Casodex®, Fugerel®, Megace®, Androcur® (no wash-out allowed)
* Previous orchiectomy, adrenalectomy or hypophysectomy
* Previous prostatic surgery (e.g. radical prostatectomy, transurethral resection of the prostate [TUR-P]) within 2 weeks of baseline
* Previous local therapy to the primary tumor with a curative attempt other than surgery (external beam radiotherapy, brachytherapy, thermotherapy, cryotherapy) within 2 weeks of baseline
* Any investigational drug within 5 half-lives of its physiological action or 3 months (whichever is longer) before baseline
* Administration of 5-alpha-reductase inhibitors (Proscar®, Avodart®, Propecia®) within 3 months before baseline
* Over-the-counter (OTC) or alternative medical therapies which have an estrogenic or anti-androgenic effect (i.e., PC-SPES, saw palmetto, Glycyrrhiza®, Urinozinc®, dehydroepiandrosterone [DHEA]) within the 3 months before baseline
* Hematological parameters (RBC, total and differential WBC count, platelet count, hemoglobin, hematocrit) outside 20% of the upper or lower limits of normal (ULN, LLN) for the clinical laboratory at screening
* Co-existent malignancy, according to the Investigator's opinion
* Uncontrolled congestive heart failure, myocardial infarction or a coronary vascular procedure (e.g. balloon angioplasty, coronary artery bypass graft) or significant symptomatic cardiovascular disease(s) within 6 months before baseline; resting uncontrolled hypertension: (>/= 160/100 mmHg) or symptomatic hypotension within 3 months before baseline
* Venous thrombosis within 6 months of baseline
* Insulin-dependent diabetes mellitus
* History of drug and/or alcohol abuse within 6 months of baseline
* Serious concomitant illness(es) or disease(s) [e.g., hematological, renal, hepatic, respiratory, endocrine, psychiatric] that may interfere with, or put patients at additional risk for, their ability to receive the treatment outlined in the protocol
* Patients receiving anticoagulants who have prothrombin and partial thromboplastin times outside of the normal range for the laboratory assays; patients who are on anticoagulation or antiplatelet medications (e.g. dipyridamole, ticlopidine, warfarin derivatives) who are not receiving a stable dose for 3 months before baseline; patients who are receiving warfarin-derivative anticoagulants who do not have an International Normalized Ratio (INR) in the therapeutic range for the clinical indication for which the anticoagulant has been prescribed.
* Blood donations/losses within 2 months of baseline, apart from previous prostatic surgery patients (see earlier exclusion [9]; please note that these patients should not be included in the pharmacokinetic [PK] group)
* Known hypersensitivity to GnRH, GnRH agonist, including any LHRH analogues, or any excipients of the study formulation
* History of the following prior to the study:

  * immunization (within 4 weeks of baseline);
  * flu shots (within 2 weeks of baseline);
  * anaphylaxis;
  * skin disease which would interfere with injection site evaluation;
  * dermatographism will be documented at screening and followed up while on treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-09; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Efficacy: to determine the proportion of patients achieving castration levels of plasma testosterone (defined as <0.5 ng/mL) 4 weeks after the first administration
to determine the proportion of patients maintaining castration levels of plasma testosterone from week 4 to study end
to determine the proportion of patients showing acute rises in plasma testosterone levels upon repeated dosing from week 4 to study end
Safety: evaluation of the safety of the new formulation based on adverse events (AEs), local tolerability, vital signs, electrocardiograms (ECGs), and clinical parameters

SECONDARY OUTCOMES:
Efficacy: determination of serum luteinizing hormone (LH), follicle-stimulating hormone (FSH), and prostate-specific antigen (PSA) concentrations
World Health Organization/Eastern Cooperative Oncology Group (WHO/ECOG) performance status, bone pain, urinary symptoms and urinary pain after administration

CONTACTS AND LOCATIONS:
Locations (28):
- United States (15):
  - Urology Centers of Alabama, Homewood, Alabama
  - Desert Oasis Cancer Center, Casa Granda, Arizona
  - Southwest Florida Urologic Associates, Fort Myers, Florida
  - Advanced Research Institute, Inc., New Port Richey, Florida
  - Florida Urology Specialists, Sarasota, Florida
  - Regional Urology, Shreveport, Louisiana
  - Lakeside Urology, Saint Joseph, Michigan
  - Hamilton Urology, P.A., Hamilton, New Jersey
  - Lawrenceville Urology, Lawrenceville, New Jersey
  - AccuMed Research Associates, Garden City, New York
  - Urological Surgeons of Long Island, Garden City, New York
  - Hudson Valley Urology, Kingston, New York
  - Hudson Valley Urology, Poughkeepsie, New York
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates, PC, Nashville, Tennessee
- Department of Urology, Vienna University Medical School, Vienna, Austria
- Czechia (4):
  - Urocentrum Praha, Prague
  - Charles University, Clinic of Urology, Prague
  - Urology Department, Hviezdoslavova, Prague
  - Masaryk Hospital, Urology Dept., Ústí nad Labem
- Department of Urology, Technical University of Dresden, Dresden, Germany
- Hungary (2):
  - Department of Urology, Semmelweis University, Budapest
  - Department of Urology, Medical School, University of Pécs, Pécs
- Italy (2):
  - Department of Urology, General Hospital of Bolzano, Bolzano
  - Sexual Medicine Unit and Urology, Università Vita Salute San Raffaele Fondazione Centro San Raffaele del Monte Tabor, Milan
- Department of Urology, Jessenius Faculty of Medicine, Comenius University, Martin, Slovakia
- Institut Català d'Oncologia, Hospital Duran I Reynals, Servicio de Oncologia Medica, Barcelona, Spain
- Royal Free Hospital and School of Medicine, London, United Kingdom

REFERENCES:
- [Derived] Marberger M, Kaisary AV, Shore ND, Karlin GS, Savulsky C, Mis R, Leuratti C, Germa JR. Effectiveness, pharmacokinetics, and safety of a new sustained-release leuprolide acetate 3.75-mg depot formulation for testosterone suppression in patients with prostate cancer: a Phase III, open-label, international multicenter study. Clin Ther. 2010 Apr;32(4):744-57. doi: 10.1016/j.clinthera.2010.04.013. PMID 20435244